CLINICAL TRIAL: NCT06983821
Title: Safe Effective Therapy With Low-Dose Glucocorticoid in ANCA-Associated Vasculitis (SAFE-LOW) Trial
Brief Title: Safe Effective Therapy With Low-Dose Glucocorticoid in ANCA-Associated Vasculitis (SAFE-LOW)
Acronym: SAFE-LOW
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250118-01T
Record Dates: First submitted 2025-04-01; First posted 2025-05-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis (MPA)
Keywords: ANCA-associated vasculitis; cyclophosphamide; glucoccorticoid; rituximab; vasculitis; granulomatosis with polyangiitis; microscopic polyangiitis; GPA; MPA
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — Cyclophosphamide; Standard of Care; Prednisone; Rituximab

STUDY DESIGN:
Intervention Model Description: Open-label, randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): IV Cyclophosphamide x 2 doses AND Rituximab AND Prednisone x 4 weeks
  Interventions: Drug: Cyclophosphamide; Drug: Prednisone; Drug: Rituximab (R)
- Standard of care (Active Comparator): Participants in this arm receive standard of care treatment induction agent and glucocorticoid dose/duration, left to the discretion of the investigator
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Drug: Cyclophosphamide — IV Cyclophosphamide 15mg/kg/dose (age and eGFR adjusted), 2 doses 2 weeks apart
  Other Names: Cytoxan
  Arms: Intervention Arm
Drug: Standard of Care (SOC) — Participants will receive standard of care induction agent and glucocorticoid taper, at investigator discretion
  Arms: Standard of care
Drug: Prednisone — 4 weeks prednisone taper
  Arms: Intervention Arm
Drug: Rituximab (R) — Rituximab infusions, dosing and schedule at clinician/investigator discretion
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a therapeutic regimen consisting of 4 weeks of glucocorticoids given with a combination of the usual induction agents for ANCA-associated vasculitis. The trial will compare this regimen to the current standard of care treatment and glucocorticoid dosing for ANCA-associated vasculitis with severe kidney involvement. This trial will begin as a pilot to assess feasibility of recruitment and of adherence to the intervention.

DETAILED DESCRIPTION:
ANCA-associated vasculitis (AAV) is an auto-immune disease which often involves the kidneys. It is a serious condition as it can lead to severe kidney impairment, often kidney failure, and may even be life-threatening. Current treatments, typically cyclophosphamide (CYC) or rituximab (RTX) with a tapering course of glucocorticoids (GC), allow most patients to achieve control of their disease (remission). Glucocorticoids are most often used initially at high doses, and then gradually decreased to low doses over at least 6 months. This leads to major treatment toxicities, notably infections and GC-related adverse events, major contributors to patient morbidity and mortality. Recent research has focused on finding ways to reduce treatment-related toxicities without compromising efficacy for controlling disease manifestations. This includes a reduced-dose GC taper for severe AAV from the Plasma Exchange and Glucocorticoids in Severe ANCA-Associated Vasculitis (PEXIVAS) trial, an even more reduced-dose GC taper in patients with moderate severity AAV from the Effect of Reduced-Dose vs High-Dose Glucocorticoids Added to Rituximab on Remission Induction in ANCA-Associated Vasculitis (LOVAS) trial, and a novel GC-sparing agent examined in the Avacopan for the Treatment of ANCA-Associated Vasculitis (ADVOCATE) trial. Despite these advances, patients still experience high rates of infections, one of the major causes of death in the first year after diagnosis, particularly in patients with most severe forms of disease. Also, novel GC-sparing drugs are costly and have limited availability throughout the world; patients who cannot access this get exposed to significant amounts of GC and must suffer their dreaded side effects.

This study addresses the unresolved issues of unacceptably high infection risk and of providing a widely available means of reducing GC exposure to minimise treatment side effects. The investigators will examine an induction treatment regimen for severe AAV consisting of 2 doses of IV CYC in combination with 4 weeks of GC and standard RTX. The control arm will be the current standard of care treatment for severe AAV. Non-controlled studies suggest the use of short duration CYC with RTX allows for minimisation of up-front GC use, as little as 1-2 weeks, but this needs to be tested in a prospective, controlled manner. The investigators hypothesize that the combination of CYC with standard RTX will allow less GC to be used for AAV. This study will begin as a pilot to examine the feasibility of the conducting the study, adherence to the intervention regimen, and of recruiting patients. If feasibility is demonstrated, the study will be extended to a full-scale trial.

ELIGIBILITY:
* New diagnosis of, or relapse of, granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA), consistent with Chapel-Hill consensus definitions
* Positive ELISA test for anti-meyloperoxidase (MPO) or anti-proteinase 3 (PR3)
* Severe kidney involvement from active AAV, characterised by both of the following:
* eGFR < 40ml/min/1.73m2 (Patients known to have a stable eGFR <40 ml/min/1.73m2 for >3 months prior to enrollment are NOT eligible)
* Biopsy proven at least focal necrotizing/crescentic glomerulonephritis OR active urinary sediment by microscopy (greater than or equal to 10 red blood cells [RBC]/high power field with erythrocyte casts or greater than or equal to 20% dysmorphic RBCs or greater than or equal to 5% acanthocytes without an alternative cause.

Exclusion Criteria (any of the following)

* A diagnosis of vasculitis other than GPA or MPA (including eosinophilic granulomatosis with polyangiitis, IgA vasculitis, cryoglobulinemic vasculitis, rheumatoid vasculitis)
* Positive anti-glomerular basement membrane antibody test or renal biopsy demonstrating linear glomerular immunoglobulin deposition
* A diagnosis of systemic lupus erythematosus or Sjögren's syndrome
* Receipt of dialysis for >21 days immediately prior to randomization or prior renal transplant
* Age <18
* Pregnant at time of screening
* Treatment with >1 IV dose of CYC and/or >14 days PO CYC and/or >14 days of prednisone/prednisone (less than or equal to 30mg/day) and/or >1 dose of RTX within the 28 days immediately prior to randomization
* Chronic viral infection: HIV. HBV or HCV
* Untreated latent mycobacterium tuberculosis infection
* Active infection at time of presentation
* A comorbidity or condition that, in the opinion of the investigator, precludes the use of GC, CYC or RTX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Pilot trial: percent adherence to intervention regimen | 12 weeks
  Pilot trial: percent adherence in the intervention arm (non-adherence will be defined as the use of more than 25% of the total expected oral prednisone in the intervention arm at 12 weeks)
Full-scale trial: Rate of serious infection | 26 weeks
  Full-scale trial: rate of serious infection (Infection occurring after randomisation requiring IV antibiotics, or leading to hospitalisation or death)

SECONDARY OUTCOMES:
Pilot trial: recruitment rate | 52 weeks
  Pilot trial: recruitment rate measured as incidence rate based on randomised participants/centre-month
Full-scale trial: Remission rate | 26 weeks
  Full-scale trial: Remission defined as absence of manifestations due to active AAV. Remission status will be determined at study visits based on clinician judgement. If a participant is not in remission at an assessment point, the affected organ system (based on Birmingham Vasculitis Activity Score [BVAS]) will be captured. If a participant is transitioned to or being planned for maintenance therapy at their study visit, then they will also be considered to have achieved remission.

OTHER OUTCOMES:
End-stage kidney disease rate | 26 and 52 weeks
  At least 12 continuous weeks of new requirement of kidney replacement therapy
Change in eGFR | 26 and 52 weeks
  Change in eGFR compared to baseline
Death | 26 and 52 weeks
  Death rate
Remission | 12, 26 and 52 weeks
  Remission rate
Rate of remission without the need for rescue therapy | 26 weeks
  Use of medications outside of the described therapies in each arm for the treatment of disease activity due to active AAV (disease flare, resistant disease or sub-optimal disease control).
Rescue therapy | 26 weeks
  Need for rescue therapy (rate)
Health-related quality of life patient-reported outcome | 4 and 12 weeks
  AAV-PRO (ANCA-associated vasculitis patient reported outcome): domain scores, scale 0-100, higher scores represent greater severity
Serious infection | 26 and 52 weeks
  Serious infection rate
Infection | 26 and 52 weeks
  Rate of infection (any severity)
Serious adverse event | 26 and 52 weeks
  Serious adverse event rate
Glucocorticoid exposure | 26 and 52 weeks
  Cumulative oral and IV prednisone equivalent dose
Weight | 12, 26 and 52 weeks
  weight change from baseline
New onset diabetes | 26 and 52 weeks
  New HbA1c >6.5%

CONTACTS AND LOCATIONS:
Overall Officials: David Massicotte-Azarniouch, MD, MSc, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - St-Joseph's Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
As per institutional requirements on protection of private health information